CLINICAL TRIAL: NCT05536115
Title: Prospective, Multicentre Clinical Trial Measuring the Impact of Treatment With ALVEOGYL in Patients With Post-extraction Dry Socket
Brief Title: Impact of Treatment With ALVEOGYL in Patients With Post-extraction Dry Socket
Status: Completed | Type: Observational
Sponsor: Septodont (Industry)
Collaborators: SMO Clinical Research (Unknown); QualityStat (Unknown)
Responsible Party: Sponsor
Other Study IDs: ALVE 2022-01; 2022-A00208-35 (Registry Identifier: ID RCB number (French)); CI/MD/2022/66273 (Registry Identifier: CI MD number (India))
Record Dates: First submitted 2022-09-07; First posted 2022-09-10 (Actual); Results first posted 2026-02-09 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-01

CONDITIONS: Dry Socket
Keywords: Tooth extraction; Dry socket; Alveolar Osteitis; Alveogyl; Surgical dressing
MeSH Terms: conditions — Dry Socket

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study population: Study patients are patients with post-extraction dry socket.
  Interventions: Device: Alveogyl

INTERVENTIONS:
Device: Alveogyl — The patients will be treated by Alveogyl. Global treatment protocol (curettage, cleaning, local anaesthesia etc.) of the dry socket is at the discretion of the Investigator.
  Alveogyl is used as an alveolar dressing. Placement of Alveogyl (about 0.2 g of paste) into the dental socket is done according to its instruction for use by a dental professional only.

SUMMARY:
Alveogyl (Septodont, Saint-Maur-des-Fossés - France) is a Medical Device used as dressing in case of dry socket.

ALVE study is a clinical investigation measuring Alveogyl performance and safety in patients with post-extraction dry socket.

The study takes place in India and in France where Alveogyl is already marketed, since 2010 in France and since 2014 in India .

ELIGIBILITY:
Inclusion Criteria:

* Male or female patient, adult or child
* Positive diagnosis of dry socket occurring after the extraction of a permanent tooth (mature or immature)
* Signed informed consent
* In France only :Patient affiliated to a Health Insurance Scheme ("sécurité sociale")

Exclusion Criteria:

* Spreading infection in the alveolar socket
* Placement of Alveogyl done immediately after tooth extraction
* Multiple post-extraction dry sockets
* Patient treated with cervico-facial radiotherapy
* Immunodeficiency related to any diseases or current treatments
* Psychiatric patient or patient unable to assess his/her pain via the study Pain VAS
* Patient with history of hypersensitivity to one of the components
* Patient on post extraction of deciduous teeth
* Participation in another clinical investigation

Min Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with a dry socket occuring after the extraction of a permanent tooth (mature or immature).
Sampling Method: Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2022-12-13 (Actual); Primary Completion 2025-06-26 (Actual); Study Completion 2025-06-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Géraldine Lescaille, DDS, PhD, Study Director — Odontology department - Pitié-Salpêtrière Hospital
Locations (16):
- France (2):
  - Hospital Henri-Mondor (AP-HP), Créteil
  - Odontology Department - Pitié-Salpêtrière Hospital, Paris
- India (14):
  - Mallige Hospital, Bangalore, Karnataka
  - Smile Dental Care, Bangalore, Karnataka
  - Perfect Dental Studio, Bangalore, Karnataka
  - Cavalier Hospital, Bangalore, Karnataka
  - Smile Dental Clinic, Bangalore, Karnataka
  - The Dental Avenues, Bangalore, Karnataka
  - Sri Dental Multispeciality Dental Hospital, Hyderabad
  - Vrisa Dental, Hyderabad
  - Eledent International Digital Dentistry, Hyderabad
  - Vardhaman Dental Care, Mumbai
  - Mayur Dental Clinic, Mumbai
  - Smile Gallery Dental Care Center, Pune
  - Dr. Salke Dental & Implant Centre, Pune
  - Sri Siddhartha Dental College, Tumakuru

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Groups:
- Study Population: Study patients are patients with post-extraction dry socket.
  Alveogyl: The patients will be treated by Alveogyl. Global treatment protocol (curettage, cleaning, local anaesthesia etc.) of the dry socket is at the discretion of the Investigator.
  Alveogyl is used as an alveolar dressing. Placement of Alveogyl (about 0.2 g of paste) into the dental socket is done according to its instruction for use by a dental professional only.
Period: Overall Study
Arm/Group | Study Population
Started | 120
Completed | 115
Not Completed | 5

BASELINE CHARACTERISTICS:
Arm/Group | Study Population
Number analyzed (Participants) | 120
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.6 (15.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 82
  Male | 38
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  France | 30
  India | 90

OUTCOME MEASURES:

1. Primary Outcome: Pain Using a Visual Analog Scale (VAS : 0-10)
Description: Patients with no pain or mild pain at Day7 The pain is measured by patients in a diary using a Visual Analogue Scale (VAS: 0-10 mm; 0 no pain - 10 maximum pain) 7 days after treatment with Alveogyl.
Time Frame: 7 days post-treatment
Population: PP Population
Measure: Count of Participants; unit: Participants
Arm/Group | Study Population
Number analyzed (Participants) | 110
Participants
  Success : Patients with no pain or mild pain at Day7 (VAS<4) | 106
  Failure : Patients with moderate to severe pain at Day 7 (VAS ≥ 4) | 4

2. Secondary Outcome: Analgesic Use
Description: Patient reporting a painkiller intake. The patient will report in a diary the intake of analgesic use at 3, 5 and 7 days after treatment with Alveogyl
Time Frame: 3 and 5 days post-treatment
Population: PP population
Measure: Count of Participants; unit: Participants
Groups:
- PP Population: Study patients are patients with post-extraction dry socket.
  Alveogyl: The patients will be treated by Alveogyl. Global treatment protocol (curettage, cleaning, local anaesthesia etc.) of the dry socket is at the discretion of the Investigator.
  Alveogyl is used as an alveolar dressing. Placement of Alveogyl (about 0.2 g of paste) into the dental socket is done according to its instruction for use by a dental professional only.
Arm/Group | PP Population
Number analyzed (Participants) | 110
Participants
  Patient reporting a painkiller intake at 3 days after treatment with Alveogyl: Patient reporting a painkiller intake | 63
  Patient reporting a painkiller intake at 3 days after treatment with Alveogyl: Patient not reporting a painkiller intake | 47
  Patients reporting a painkiller intake at 5 days after treatment with Alveogyl: Patient reporting a painkiller intake | 20
  Patients reporting a painkiller intake at 5 days after treatment with Alveogyl: Patient not reporting a painkiller intake | 90

3. Secondary Outcome: Healing of the Alveolar Mucosa
Description: Healing of the alveolar mucosa will be clinically reported by the dentist using le Wound healing index.
  The Wound Healing Index ranges from 1 (poor healing) to 5 (excellent healing), with higher scores indicating better gingival wound healing.
Time Frame: 7 days post-treatment
Measure: Mean (Standard Deviation); unit: Wound healing index Score
Arm/Group | Study Population
Number analyzed (Participants) | 110
Wound healing index Score | 4.0 (0.8)

4. Secondary Outcome: Signs of Local Inflammation
Description: Signs of inflammation around the gingival mucosa (oedema, redness, sensitivity) will be reported by the dentist at Day 7 after tratment with Alveogyl
Time Frame: 7 days post-treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Study Population
Number analyzed (Participants) | 110
Participants
  patients showing signs of inflammation around the gingival mucosa | 19
  patients without signs of inflammation around the gingival mucosa | 91

5. Secondary Outcome: Antiseptic Effect
Description: Any clinical signs such as gum pain, swollen gum lining, fever, halitosis,...) will be reported by the dentist
Time Frame: 7 days post-treatment
Population: PP population
Measure: Count of Participants; unit: Participants
Arm/Group | Study Population
Number analyzed (Participants) | 110
Participants
  Halitosis / bad breath: Yes | 12
  Halitosis / bad breath: No | 96
  Halitosis / bad breath: Unknown | 2
  Fever: Yes | 2
  Fever: No | 108
  Fever: Unknown | 0
  Tenderness of the gingival mucosa: Yes | 24
  Tenderness of the gingival mucosa: No | 86
  Tenderness of the gingival mucosa: Unknown | 0
  Purulent collection in the alveolus and gingival mucosa: Yes | 0
  Purulent collection in the alveolus and gingival mucosa: No | 110
  Purulent collection in the alveolus and gingival mucosa: Unknown | 0
  Pale discoloration of the dry socket: Yes | 17
  Pale discoloration of the dry socket: No | 93
  Pale discoloration of the dry socket: Unknown | 0

6. Secondary Outcome: Hemostasis
Description: Presence or absence of bleeding in the socket.
Time Frame: Immediately after Alveogyl placement and Day 7 after treatment
Population: PP population
Measure: Count of Participants; unit: Participants
Arm/Group | Study Population
Number analyzed (Participants) | 110
Participants
  Presence or absence of bleeding in the socket immediately after Alveogyl placement: Patients without Bleeding | 96
  Presence or absence of bleeding in the socket immediately after Alveogyl placement: Patients showing mild bleeding | 13
  Presence or absence of bleeding in the socket immediately after Alveogyl placement: Patients showing moderate bleeding | 1
  Presence or absence of bleeding in the socket immediately after Alveogyl placement: Patients showing hemorrhagic oozing | 0
  Presence or absence of bleeding in the socket 7 days after Alveogyl placement: Patients without Bleeding | 110
  Presence or absence of bleeding in the socket 7 days after Alveogyl placement: Patients showing mild bleeding | 0
  Presence or absence of bleeding in the socket 7 days after Alveogyl placement: Patients showing moderate bleeding | 0
  Presence or absence of bleeding in the socket 7 days after Alveogyl placement: Patients showing hemorrhagic oozing | 0

7. Secondary Outcome: Complication Rate
Description: Adverse events occuring within 7 days after treatment
Time Frame: From Alveogyl placement to 7 days post-treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Study Population
Number analyzed (Participants) | 110
Participants
  Patients with adverse events | 0
  Patients without adverse events | 110

ADVERSE EVENTS:
Time Frame: 7 days
Arm/Group | Study Population
All-Cause Mortality (participants affected / at risk) | 0/120
Serious Adverse Events (participants affected / at risk) | 0/120
Other Adverse Events (participants affected / at risk) | 0/120

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-01-22): https://cdn.clinicaltrials.gov/large-docs/15/NCT05536115/Prot_SAP_000.pdf